CLINICAL TRIAL: NCT03620695
Title: Probe-based Confocal Laser Endomicroscopy With Topical Cresyl Violet for Diagnosis of Colorectal Polyps
Brief Title: Confocal Laser Endomicroscopy With Topical Cresyl Violet for Colorectal Polyps
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2018SDU-QILU-03
Record Dates: First submitted 2018-07-31; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Probe-based confocal laser endomicroscopy (pCLE) has been shown to a reliable diagnostic method enabling in vivo microscopic imaging during ongoing endoscopy. Usually fluorescein then serves as a contrast agent for pCLE, but it does not allow direct nuclear visualization, must be injected, leads to a transient skin discoloration, and may have allergic side effects. This study aimed to establish a single topical dye, cresyl violet (CV) for pCLE imaging, to describe pCLE interpretation criteria for the characterization of colorectal polyps with histopathological correlation, and to perform the validation of these criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 75 years, with polyps found during surveillance or screening colonoscopies.

Exclusion Criteria:

* Contraindications to CV (such as allergy);
* Pregnancy or breastfeeding;
* Serous cardiopulmonary diseases, severe coagulopathy dysfunction, impaired kidney function;
* Inability to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients undergoing surveillance or screening colonoscopies will be recruited in this study at Qilu Hospital, Shandong University.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
The pCLE with topical CV interpretation criteria for the characterization of colorectal polyps with histopathological correlation | 5 months
Number of diagnostic agreement between pCLE with topical CV and histopathological results | 5 months
Number of participants with procedure-related adverse events | 5 months
Number of pCLE imaging failure with topical CV | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China